CLINICAL TRIAL: NCT02090387
Title: Evaluation of a Complete Oral Nutritional Supplement on Lean Body Mass in Healthy Older Subjects During Bed Rest and Recovery.
Brief Title: Evaluation of an Oral Nutritional Supplement on Lean Body Mass in Healthy Older Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: BL20; NCT02238600 (obsolete NCT alias)
Record Dates: First submitted 2014-03-17; First posted 2014-03-18 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control ONS (Active Comparator): ONS without AN777
  Interventions: Other: ONS without AN777
- Investigational ONS (Experimental): ONS containing AN777
  Interventions: Other: ONS containing AN777

INTERVENTIONS:
Other: ONS without AN777 — 2 servings a day
  Other Names: Commercially available ONS
  Arms: Control ONS
Other: ONS containing AN777 — 2 servings a day
  Other Names: Investigational ONS
  Arms: Investigational ONS

SUMMARY:
The study will evaluate the effects of oral nutritional supplements (ONS) on attenuating the lean body mass (LBM) loss that occurs after bed rest.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 to ≤ 79 years
2. Body Mass Index (BMI) >20 but ≤ 35 kg/m2.
3. Short Physical Performance Battery (SPPB) score of > 9 (fully functional with no mobility limitations).
4. Triacylglyceride (TAG) level is ≤ 250 mg/dl, LDL cholesterol is ≤ 155 mg/dl, total cholesterol level is ≤ 250 mg/dl.
5. Compliance with the various activity levels required for this study.
6. Ankle brachial index within the normal range, between 1 and 1.4.
7. Physical activity score within the 2008 Guidelines for Americans.
8. Normal-good handgrip strength.

Exclusion Criteria:

1. Type I or Type II Diabetes Mellitus.
2. Fasting blood glucose level of >115 mg/dl.
3. Major surgery, less than 6 weeks prior to enrollment in the study, or subject has planned elective surgery requiring 2 or more days of hospitalization.
4. History of pressure ulcers.
5. Stated history of Deep Vein Thrombosis (DVT), recent elevated D-dimer test, a positive ultrasound for DVT, pulmonary embolism, carotid atherosclerosis, transient ischemic attack (TIA), or stated hypercoaguable condition, or other clotting or bleeding disorders, or is currently prescribed blood thinners.
6. Varicose veins that would result in significant discomfort while wearing TED hose and/or SCD.
7. Stated autoimmune disease or active malignant disease.
8. Estimated glomerular filtration rate is < 50ml/min/1.73m2.
9. Current significantly impaired liver function or hepatic enzyme tests are ≥2.5 times normal limit.
10. Significant cardiovascular event ≤ 6 months prior to screening visit; or stated history of congestive heart failure.
11. Untreated hypo- or hyper-thyroidism, or other endocrinopathies associated with excessive androgen secretion.
12. Refractory anemia with hemoglobin value <11.0 g/dl.
13. Chronic, contagious, infectious disease, such as active tuberculosis, hepatitis B or C, or HIV.
14. Current infection (requiring prescription antimicrobial or antiviral medication, or hospitalization), or has received corticosteroid treatment (with the exception of inhaled or topical steroids) in the last 3 months.
15. Currently being prescribed pain/anti-inflammatory medication and/or is regularly consuming over the counter pain/anti-inflammatory medication for chronic, or persistent, pain, including but not limited to arthritic conditions, fibromyalgia, and continuous localized pain.
16. History of allergy to any of the ingredients in the study products.
17. Deleted
18. Obstruction of the gastrointestinal tract precluding ingestion of the study product, inflammatory bowel disease, short bowel syndrome or other severe forms of gastrointestinal disease.
19. Stated uncontrolled severe diarrhea, nausea or vomiting.
20. Amputee.
21. Actively pursuing weight loss or gain.
22. Cannot refrain from taking medications/dietary supplements (all forms)/substances that could modulate metabolism or body weight.
23. Cannot refrain from taking long chain n-3 polyunsaturated fatty acids (PUFA) (eicosapentaenoic acid (EPA) ± docosahexaenoic acid (DHA) ± α-linolenic acid (ALA)), or vitamin D, at levels that are significantly higher than the established Acceptable Macronutrient Distribution Range (AMDR), or recommended by the American Heart Association (500 mg/d total EPA+DHA), during the study.
24. Cannot refrain from smoking or discontinue the use of nicotine (all forms including patches) or tobacco during the study.
25. One or more metal implants.
26. Currently diagnosis or a history of severe dementia or delirium, eating disorder, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance.
27. Cannot abstain from alcohol use during the study.

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Total lean body mass | Baseline to Study Day 10
  Change from baseline

SECONDARY OUTCOMES:
Hand-grip strength | Baseline, Study Day 10, Study Week 6 and 12
  Change from baseline
Short Physical Performance Battery (SPPB) | Baseline, Study Day 10, Study Week 6 and 12
  Change from baseline
Isokinetic leg strength | Baseline, Study Day 10 and Study Week 12
  Change from baseline
Body Mass Index (BMI) | Screening Visits 1 and 3; Baseline; Study Days 2, 4, 6, 8 and 10; Study Weeks 3, 6, 9 and 12
  Calculated BMI = weight/height2 (kg/m2).
Lower extremity lean mass | Baseline, Study Day 10, Study Weeks 6 and 12
  Measured by DXA; Change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Owen Kelly, Ph.D, Study Chair — Abbott Nutrition
Locations (3):
- United States (3):
  - University of Arkansas for Medical Sciences (UAMS), Little Rock, Arkansas
  - Florida Hospital Translational Research Institute for Metabolism and Diabetes, Orlando, Florida
  - Center of Translational Research in Aging & Longevity, College Station, Texas

IPD SHARING:
Plan to Share IPD: Undecided